CLINICAL TRIAL: NCT04804280
Title: Epigenetics and Protective Factors in the Preterm Infant: Neural and Methylation Correlates of Developmental Care During Neonatal Intensive Care Unit Hospitalization
Brief Title: Epigenetics and Protective Factors in the Preterm Infant
Acronym: EPIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: RC2020_751
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Preterm Birth; Parent-Child Relations; Epigenetics
Keywords: At-risk Infants; Developmental Care; DNA methylation; affectionate touch; Insular cortex
MeSH Terms: conditions — Premature Birth | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will investigate the methylation status of target genes (such as BDNF, SLC6A4, OXTR, NR3C1) in preterm children (PT), compared with a sample of full term children (FT). Cord blood will be collected at birth for both PT and FT groups and, only for PT infants, a peripheral blood sample will be collected at hospital discharge, following routine clinical procedures. Blood samples will be obtained by trained nurses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm children (PT): * gestational age at birth: 26+0 to 31+6 weeks;
  * absence of documented neurological pathology;
  * absence of sensory deficits;
  * absence of malformative syndromes and/or major malformations.
  Interventions: Genetic: DNA methylation of target genes; Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI) acquisition
- Full-term children (FT): * gestational age at birth ≥ 37 weeks;
  * birth weight ≥ 2,500g;
  * APGAR 5' ≥ 7
  * delivery without any complications for baby and/or mother;
  * no prenatal and/or postnatal clinical conditions;
  * no hospitalizations at the time of birth or postpartum;
  * absence of malformative syndromes and/or major malformations.
  Interventions: Genetic: DNA methylation of target genes; Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI) acquisition

INTERVENTIONS:
Genetic: DNA methylation of target genes — The methylation status of target genes (BDNF, SLC6A4, OXTR, NR3C1) will be investigated. Cord blood will be collected at birth for PT and FT, only for PT a peripheral blood sample will be collected at hospital discharge, during routine clinical procedures. Genomic DNA will be extracted from aliquots of 0. 2 ml of each blood sample with the GeneElute Blood Genomic DNA kit (Sigma) and stored at -20°C. Aliquots of 250 ng of each DNA will be edited for methylation analysis with the EZ DNA Methylation Lightning kit (Zymo Research). Amplification of samples and their preparation for NGS sequencing will be performed. Samples will be sequenced on NextSeq 500 (Illumina). Individual processed sequences (PE reads) will be independently aligned to reference sequences using a parallel Smith-Waterman algorithm. Only reads that consistently align to the same reference sequence will be retained. At each CpG site in each analyzed sequence, the frequencies of the four bases will be evaluated.
Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI) acquisition — Infants will undergo an MRI exam with a 3 Tesla Philips Achieva scanner and a 32-channel head coil. a trained experimenter will apply tactile stimulation associated with affective touch characteristics to the child with a soft brush on the right anterior tibial region in proximal and distal directions. The length of the stimulated area will be measured to cover approximately 15 cm, and tactile stimulations will be applied at a rate of 5 cm/s for 15s, with randomized intervals between stimuli of 10-15s (resulting in 5 stimulations in a 15s block). A regular audio signal will help the researcher to keep a constant stroke velocity. Audio commands will also be used to direct the experimenter. Infant must be asleep (natural sleep) during the fMRI acquisition.

SUMMARY:
Preterm infants (PT) spend their first weeks of life in the Neonatal Intensive Care Unit (NICU) where they are exposed to unfavorable conditions with different effects on child development including long-term alterations in epigenetic regulation (DNA methylation). Recent studies document that these epigenetic changes are associated with behavioral modifications, such as altered stress reactivity at 3 months and 4 years. A growing number of studies suggest that protective Developmental Care (DC) procedures (e.g., breastfeeding, skin-to-skin contact (SSC), maternal holding) positively impact neurophysiological and behavioral adaptation of PT with long-term effects. Additionally, a neuro-imaging study reported that parental support in the NICU is associated with improved brain connectivity. While in term (FT) infants, parental interpersonal touch (breastfeeding, affectionate touch) is associated with reduced methylation and activation of specific brain areas associated with affective interpersonal touch, to date no study has investigated whether DC practices and maternal care in NICU (specifically, SSC) buffer methylation and support the brain response to affectionate physical touch in PT. The present study investigates the association between DC procedures in NICU, DNA methylation, and brain responses to affectionate touch, investigated through the use of MRI, at 2 months of age (corrected for prematurity), controlling for: (1) birth status (PT vs FT); (2) the duration of SSC during the NICU stay; (3) parental affectionate touch in the home environment and during mother-child interaction.

DETAILED DESCRIPTION:
Background: preterm infants (PT) spend their first weeks of life in the Neonatal Intensive Care Unit (NICU) where they are exposed to conditions with different effects on child development including long-term alterations in epigenetic regulation. Recent studies document that these epigenetic changes are associated with behavioral modifications, such as altered stress reactivity at 3 months and 4 years. A growing number of studies suggest that protective Developmental Care (DC) procedures (e.g., breastfeeding, skin-to-skin contact (SSC), maternal containment) positively impact neurophysiological and behavioral adaptation of PTs with long-term effects. Moreover, structural factors of the NICU, such as the organization of the unit space based on Open-Bay rather than Single Family Rooms could impact the child's neurobehavioral development and the parent's well-being. For example, a study on the impact of the Single Family Room shows improved medical and neurobehavioral outcomes for the infant at discharge and increased maternal involvement. However, the Single Family Room literature also reports mixed results with some studies finding increased parent involvement but no effect on child growth and some showing increased parent stress.

Primary aim: to evaluate the methylation status of target genes (e.g., BDNF, SLC6A4, OXTR, NR3C1) in association with exposures to DC practices during NICU hospitalization in PT children, compared with a sample of FT children.

Secondary aim: to investigate the relationship between preterm/term birth, DC practices (PT only), maternal touch in the postnatal period, epigenetic status and brain response to soft/soft stimulation during fMRI, at 2 months of age (corrected for prematurity in PT children), controlling for characteristics of the NICU of provenance (NICU Hospital of Monza: Single Family Room vs NICU Hospital of Lecco: Open-Bay).

Planned Activities:

Methods

The project is characterized as observational, micro-longitudinal and is structured in two phases:

- PHASE 1: FROM BIRTH TO DISCHARGE FOR PT CHILDREN; TIME OF BIRTH FOR FT CHILDREN)

At the time of birth, both PT and FT will have their cord blood collected (methylation at birth) using non-invasive methods. Only for PTs at the time of discharge will be performed a second blood draw at the same time as the routine pre-discharge checks. In addition, at this stage, the mother will fill out some questionnaires about her mood and will be obtained information on pregnancy and childbirth (gestational age, birth weight, length and head circumference of the child at birth, type of delivery, duration of hospitalization, presence of perinatal diseases) and socio-anagraphic variables. Finally, only for the PT group, during hospitalization in the NICU, the following data will be collected on the negative and positive experiences to which PTs are exposed during hospitalization, specifically:

1. number of pain-related stress procedures (e.g.: number of withdrawals, central insertions, invasive and non-invasive mechanical ventilation) obtained from the patient's medical record;
2. time spent doing DC procedures (e.g.:, total time spent in which the child is attached to the mother's breast, total time spent in holding, total time spent in kangaroo care) obtained through the use of the "closeness diary" implemented in electronic format, in the form of an APP.

At the end of the NICU admission, only for PT children, a second peripheral blood sampling (methylation at discharge) will be performed at the same time as routine pre-discharge checks. At the end of hospitalization, mothers of PTs will complete the same questionnaires completed at birth and in addition will be asked to complete questionnaires on the experience of stress and support received from staff during hospitalization in the NICU.

- PHASE 2: AROUND 2 MONTHS OF AGE OF THE CHILD (CORRECTED AGE FOR PT) The children of both groups (PT and FT) and their mothers will go to the IRCCS "E. Medea" for a Functional Magnetic Resonance Imaging (fMRI) examination. The fMRI session will be conducted according to a recent study on the neural correlates of maternal affective touch in FT infants. The fMRI scan will be conducted by researchers and clinicians experienced in the use of MRI in pediatric settings. Prior to the fMRI session, all parents will be adequately briefed with respect to the MRI-related procedure and the scanning protocol will be viewed with the parents and staff will confirm the absence of safety risks. To minimize the potential risk and harm to infants caused by unnecessary sedation, fMRI will be performed during natural sleep and no sedation will be performed. Infants will be wrapped, fed, and scanned. To promote falling asleep, infants will be changed and fed by their mother and given time for them to fall asleep and then moved into the scanner. All infants will be fitted with hearing protection. In the event that the infant wakes up during the scan, the mother will be asked to attempt to put the infant back to sleep and if this occurs, the scan will be attempted again. Standard hearing protection will be given to the parents who will be allowed to remain in the scanning room for the duration of the acquisition session. The scan will be observed by control room staff. The entire procedure was structured in accordance with the guidelines for conducting fMRI in healthy child samples. After the fMRI, a 10-minute video recording of the mother-child interaction will be made. During the video recording, the child will be placed in a comfortable infant seat and the mother will be asked to sit in front of the child and interact with him/her for 5 min. Baby and mother's behavior and interaction will be coded using the Global Rating Scales mother-child interaction coding system and maternal touch coding using the Maternal Touch Coding System.

ELIGIBILITY:
Inclusion criteria for PT children are:

* gestational age: 26+0 to 31+6 weeks;
* absence of documented neurological pathology;
* absence of sensory deficits;
* absence of malformative syndromes and/or major malformations.

Inclusion criteria for FT infants are:

* gestational age ≥ 37weeks;
* birth weight ≥ 2,500g;
* APGAR 5' ≥ 7 - delivery without any complications for the child and/or mother;
* no pre/postnatal/postnatal clinical conditions;
* no hospitalizations at the time of birth or postpartum;
* absence of malformative syndromes and/or major malformations.

Inclusion criteria for mothers are:

* mothers of Italian nationality;
* mother over 18 years of age;
* mother with absence of manifest psychiatric and/or cognitive pathologies (must be previously diagnosed major psychiatric pathologies);
* non-addicted/no habitual use of psychotropic medications, drugs, alcohol no smoking;
* non-single-parent families.

Exclusion criteria: refer to inclusion criteria.

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants. Preterm infants infants will be pre-screened for medical status variables by the NICU neonatologists of different hospital in Lombardy. Following a letter outlining the general research, parents will be meet per person in NICU or contacted by telephone and asked to voluntarily participate.
  Full-term infants. Mothers and their infants will be enrolled during the prenatal/ postnatal parenting coursein different hospital in Lombardy. Following a letter outlining the general research, parents will be contacted by telephone and asked to voluntarily participate.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-04-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
DNA methylation changes in PT | first 6 months (Corrected Age for PT) of infant's life
  Correlation between DNA methylation changes of target genes (BDNF, SLC6A4, OXTR, NR3C1) and the duration of Developmental Care practice that involved proximity and pyisical contact during the NICU stay measured by a specific APP.

SECONDARY OUTCOMES:
Insular cortex and somatosensory cortex activation in PT and FT infants | when the infants is 2 months-old (Corrected Age for PT)
  Significant differences in mean BOLD signal magnitude in the insular cortex and in somatosensory cortex between PT and FT in the slow skin stroking experimental task during the fMRI session.
Developmental Care procedures in NICU and insular cortex/somatosensory cortex activation in preterm infants | first 2 months (Corrected Age for PT) of infant's life
  Correlation between the duration of Developmental Care practice taht involved proximity and physical contact during the NICU stay measured by a specific APP and mean BOLD signal magnitude in the insular cortex and in somatosensory cortex (in the slow skin stroking experimental task during the fMRI session) in PT.

CONTACTS AND LOCATIONS:
Locations (1):
- Associalzione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy